CLINICAL TRIAL: NCT00129311
Title: Usefulness of Selegiline for Smoking Cessation
Brief Title: Usefulness of Selegiline as an Aid to Quit Smoking - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA-15757-1; R01DA015757 (NIH); R01-15757-1; DPMC
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Results first posted 2014-07-16 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2014-07

CONDITIONS: Tobacco Use Cessation
Keywords: Tobacco
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Selegiline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Selegiline
  Interventions: Drug: Selegiline
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Selegiline — 5 mg capsules taken by mouth. Participants take 5 mg once a day for the first week of the study, then increase the dose to 5 mg twice a day for 6 weeks, then take 5 mg once a day during the last week of the study. Participants receiving the placebo pill take 1 pill per day for the first week of the study and 1 pill twice a day for the other weeks.
  Other Names: L-deprenyl; Eldepryl®
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
Despite the widespread use of nicotine replacement therapies for the treatment of nicotine dependence, many smokers are still unable to quit smoking. The purpose of this study is to determine the safety and effectiveness of selegiline as an aid to help smokers quit smoking.

DETAILED DESCRIPTION:
Despite the availability of nicotine replacement therapies and sustained-relapse bupropion for the treatment of nicotine dependence, there is still a significant proportion of cigarette smokers who are unable to quit smoking. Therefore, new and effective pharmacotherapies for smoking cessation are needed. The primary aim of this study is to determine the safety and efficacy of selegiline as an aid to smoking cessation.

In this study, 200 nicotine-dependent cigarette smokers will participate in an 8-week, double-blind, placebo-controlled trial and then will be followed over 4 years. Participants will be randomly assigned to receive either selegiline or placebo. Selegiline doses of 5 mg will be taken once a day during the first week. This will be increased to 5 mg twice daily for the remaining 7 weeks. The target smoking "quit date" will be Day 15. All smokers will receive brief weekly manualized smoking cessation counseling from the Mayo Clinic's "Smoke Free and Livin' It" program. The primary smoking cessation outcome measure will be 7-day point prevalence smoking abstinence at the 6-month follow-up. Secondary cessation outcome measures will include continuous smoking abstinence during the last four weeks of the trial (Days 29-56) and 7-day point prevalence abstinence at the end of the 8-week trial (Days 49-56).

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for nicotine dependence with a Fagerstrom Test of Nicotine Dependence (FTND) score greater than 5
* Smokes at least 15 cigarettes daily (averaged over 1 week, within the month prior to enrollment)
* Motivated to quit smoking within 30 days at time of initial evaluation
* At least one unsuccessful attempt to quit smoking in the past year
* An expired breath CO level greater than 10 ppm and baseline plasma cotinine level greater than 150 ng/ml at initial evaluation
* Body weight of at least 100 lb
* Avoidance of nicotine replacement product use one month prior to enrollment
* Speaks English

Exclusion Criteria:

* Currently taking over-the-counter or prescription sympathomimetic agents (e.g., pseudoephedrine, methylphenidate), antidepressant agents (e.g., tricyclic antidepressants, serotonin reuptake inhibitors, bupropion, other monoamine oxidase inhibitors), or meperidine (Demerol)
* Serious medical disorders such as unstable angina or liver failure
* Abnormalities in baseline bloodwork (e.g., threefold elevation of liver function tests, electrolyte abnormalities)
* Physiologically dependent on and/or abusing alcohol or other drugs of abuse (e.g., cocaine, opiates, benzodiazepines, etc.) during the 6 months prior to enrollment (based on a clinical evaluation, which includes a self-report, and is confirmed by a positive urine toxicology screen)
* Meets DSM-IV criteria for a current diagnosis of major depressive disorder, panic disorder, or post-traumatic stress disorder
* Current or past history of bipolar disorder or schizophrenia
* Past history of major depression associated with historical evidence of suicidal or homicidal behavior, or psychotic symptoms
* Currently residing with another study participant
* Presence of suicidal or homicidal ideation
* Significant impairment of social or occupational functioning, either at time of initial evaluation or during the trial
* Known hypersensitivity to selegiline hydrochloride

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2004-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony P George, M.D., Principal Investigator — Yale University; Marc N Potenza, M.D., Ph.D., Principal Investigator — Yale University
Locations (1):
- PRISM, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961
- [Derived] Weinberger AH, Reutenauer EL, Jatlow PI, O'Malley SS, Potenza MN, George TP. A double-blind, placebo-controlled, randomized clinical trial of oral selegiline hydrochloride for smoking cessation in nicotine-dependent cigarette smokers. Drug Alcohol Depend. 2010 Mar 1;107(2-3):188-95. doi: 10.1016/j.drugalcdep.2009.10.009. Epub 2009 Nov 24. PMID 19939587

RESULTS

PARTICIPANT FLOW:
Groups:
- Selegiline: Selegiline
  Selegiline: 5 mg capsules taken by mouth. Participants take 5 mg once a day for the first week of the study, then increase the dose to 5 mg twice a day for 6 weeks, then take 5 mg once a day during the last week of the study. Participants receiving the placebo pill take 1 pill per day for the first week of the study and 1 pill twice a day for the other weeks.
- Placebo: Placebo
  Selegiline: 5 mg capsules taken by mouth. Participants take 5 mg once a day for the first week of the study, then increase the dose to 5 mg twice a day for 6 weeks, then take 5 mg once a day during the last week of the study. Participants receiving the placebo pill take 1 pill per day for the first week of the study and 1 pill twice a day for the other weeks.
Period: Overall Study
Arm/Group | Selegiline | Placebo
Started | 51 | 50
Completed | 39 | 31
Not Completed | 12 | 19
Not completed — Withdrawal by Subject | 12 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Selegiline | Placebo | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (11.0) | 46.2 (13.0) | 47.4 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 26 | 24 | 50
Region of Enrollment [Number; unit: participants]
  United States | 51 | 50 | 101
Education [Mean (Standard Deviation); unit: years] | 13.8 (2.0) | 14.2 (2.2) | 14.0 (2.1)
Age of Smoking Onset [Mean (Standard Deviation); unit: years] | 16.2 (6.9) | 16.3 (4.1) | 16.3 (5.6)
Duration of Smoking (years) [Mean (Standard Deviation); unit: years] | 31.6 (11.6) | 29.8 (13.6) | 30.7 (12.6)

OUTCOME MEASURES:

1. Primary Outcome: 7 Day Point Prevalence of Cigarette Abstinence
Time Frame: 6-month follow up
Measure: Number; unit: participants
Arm/Group | Selegiline | Placebo
Number analyzed (Participants) | 51 | 50
participants | 6 | 8

2. Primary Outcome: 7 Day Point Prevalence of Cigarette Abstinence
Time Frame: Week 8
Measure: Number; unit: participants
Arm/Group | Selegiline | Placebo
Number analyzed (Participants) | 51 | 50
participants | 8 | 10

ADVERSE EVENTS:
Arm/Group | Selegiline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50
Other Adverse Events (participants affected / at risk) | 47/51 | 45/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selegiline (N=51) | Placebo (N=50)
Dry Mouth (General disorders) | 13 | 4
Flu Like Symptoms (General disorders) | 11 | 4
Irregular or Rapid Heartbeat (General disorders) | 9 | 5
Headaches (General disorders) | 24 | 21
Drowsiness (General disorders) | 20 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No